CLINICAL TRIAL: NCT02471417
Title: Dietary Nitrate Supplementation in Dilated Cardiomyopathy: An Acute, Double-blind, Randomized, Placebo-controlled, Crossover Trial.
Brief Title: Acute Dietary Nitrate in Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University College Dublin (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Acute NO3- in DCM
Record Dates: First submitted 2015-01-07; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental): Concentrated, beetroot juice is a rich source of dietary nitrate.
  Interventions: Dietary Supplement: Dietary nitrate
- Nitrate depleted placebo beetroot juice (Placebo Comparator): Placebo beetroot juice is identical to active beetroot juice in every way except nitrate content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary nitrate — 140ml of nitrate rich beetroot juice provides 12.9mmol nitrate and will be on a single occasion by the study subjects.
  Other Names: Beetroot juice
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Placebo — 140ml of nitrate depleted beetroot juice provides 0.5mmol nitrate and will be on a single occasion by the study subjects.
  Other Names: Nitrate depleted beetroot juice
  Arms: Nitrate depleted placebo beetroot juice

SUMMARY:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to improve exercise capacity in athletes, healthy adults and subjects with both peripheral vascular disease or COPD. Many patients with dilated cardiomyopathy have reduced exercise capacity, The investigators hypothesized that acute nitrate consumption might increase incremental shuttle walk test (ISWT) distance in dilated cardiomyopathy subjects compared to a placebo beetroot juice.

DETAILED DESCRIPTION:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to improve exercise capacity in athletes, healthy adults and subjects with both peripheral vascular disease or COPD. Many patients with dilated cardiomyopathy have reduced exercise capacity, The investigators hypothesized that acute nitrate consumption might increase incremental shuttle walk test (ISWT) distance in dilated cardiomyopathy subjects compared to a placebo beetroot juice. This study is a randomized, double-blind placebo-controlled, crossover trial. Resting blood pressure, phlebotomy and ISWT will be performed. Following completion, each subject is randomized to consume beetroot juice or placebo. 3 hours later, the same assessments are repeated by the same people. After a 7d washout, the entire protocol is repeated with the crossover beverage.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable,
* Confirmed non-ischemic, dilated cardiomyopathy

Exclusion Criteria:

* Active musculo-skeletal conditions
* Ischemic heart disease
* Pulmonary hypertension
* COPD
* Taking vasodilators
* Diabetes mellitus

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change between incremental shuttle walk test distance pre and post juice | Day 1 and day 8

SECONDARY OUTCOMES:
Clinic blood pressure | Day 1 and day 8
Plasma nitrate | Day 1 and day 8
Dyspnoea using self report, validated Borg scale | Day 1 and day 8
Oxygen saturation using pulse oximetry | Day 1 and day 8
Plasma nitrite | Day 1 and day 8

CONTACTS AND LOCATIONS:
Overall Officials: Jim O 'Neill, MD, Principal Investigator — Connolly Hospital Blanchardstown